CLINICAL TRIAL: NCT05709561
Title: The Effect of Acupressure and Mindfulness to Cope With Premenstrual Syndrome on Premenstrual Symptoms and Quality of Life
Brief Title: The Effect of Acupressure and Mindfulness to Cope With Premenstrual Syndrome (PMS) on PMS and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Simge Ozturk, Pricipal Investigator, Inonu University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2022/3172
Record Dates: First submitted 2022-12-25; First posted 2023-02-02 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Premenstrual Syndrome
Keywords: Acupressure; Mındfulness; Nurse; Quality of life
MeSH Terms: conditions — Premenstrual Syndrome | interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant
Masking Description: Student
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acupressure Group (Active Comparator): Acupressure was applied to the acupressure group twice a week in the first week by the researcher. Then, in the second week, it was observed that the students themselves applied this application twice this week under the supervision of the researcher.Then the acupressure group was asked to apply acupressure two days a week for 12 weeks, a total of 24 times.
  Interventions: Procedure: Acupresur
- Mindfulness Group (Active Comparator): The researcher and students practiced mindfulness once a week for 8 weeks. Then the students were asked to do 3 cycles of application alone every day. mid-test was applied.
  Interventions: Procedure: Mindfulness
- Plasebo Group (Placebo Comparator): Acupressure and mindfulness practices were not applied to the control group and they continued their routine care.
  Interventions: Procedure: Plasebo

INTERVENTIONS:
Procedure: Acupresur — acupressure application was applied 2 times a week for a total of 12 weeks and 24 times.
  Arms: Acupressure Group
Procedure: Mindfulness — Mindfulness practice was applied with the students once a week for 8 weeks, accompanied by a researcher. Then, students were asked to apply for 3 cycles.
  Arms: Mindfulness Group
Procedure: Plasebo — No intervention was applied to the control group.
  Arms: Plasebo Group

SUMMARY:
The research was carried out to determine the effect of acupressure and mindfulness practice to cope with premenstrual syndrome on premenstrual symptoms and quality of life. The sample of the study consisted of a total of 270 students, 90 of which were acupressure, 90 mindfulness and 90 control groups. In the study, data were collected with the Participant Information Form, PMSS and WHOQOL-BREF. The acupressure group was asked to apply acupressure two days a week for 12 weeks, a total of 24 times. In the mindfulness group, 8 weeks of Conscious Awareness Stress Reduction Program was applied, after which the students were asked to practice mindfulness for 3 cycles. Students in both experimental groups were asked to stop the practices after acupressure and mindfulness practices. PMSS and WHOQOL-BREF were applied to both experimental and control groups as an intermediate test 12 weeks after the pre-test and a post-test 24 weeks later.

DETAILED DESCRIPTION:
Premenstrual syndrome (PMS) is a gynecological condition consisting of physical, psychological and behavioral symptoms that occur 7-10 days before menstruation and end with the onset of menstruation. Symptoms are divided into three groups as mild, moderate and severe. The prevalence of PMS is reported to be 47.8% on average worldwide. About 20% of these are severe symptoms and may affect women's daily activities, while 27.8% are mild to moderate symptoms. PMS reduces daily activities, sleep quality and cognitive functions of women of reproductive age. However, it can negatively affect women's health, interpersonal relationships, academic performance, attendance at work and school, and quality of life. In the treatment of PMS, 80% of women prefer non-pharmacological treatment. Non-pharmacological methods such as lifestyle changes, music, massage, yoga, aromatherapy, reflexology, homeopathy, cognitive behavioral therapy, emotional liberation technique, reiki, acupuncture, mindfulness, acupressure methods are frequently used in the treatment of PMS. The population of the research consists of 1006 female students, 598 of whom are studying at İnönü University Faculty of Nursing and 408 female students studying at Bartın University Faculty of Health Sciences. The sample of the study was determined by power analysis with an effect size of 0.22, a confidence interval of 0.95 determined by an error level of 0.05, a sample size of 90 for each group (90 in the acupressure group, 90 in the mindfulness group, and 90 in the control group) with 0.95 universe representation power. group 90) female students with a total of 270 PMS were determined. However, it was decided to include an additional 10 students for each group, taking into account the losses that may occur during the study. In the study, 100 acupressure, 100 mindfulness and 100 female students formed the control group. In the study, which university would be included in the control and experimental groups was determined by drawing lots. The draw was made blind by an academic independent of the research. As a result of the lottery, the control group of the research was formed by the students of İnönü University Faculty of Nursing, and the experimental groups were students studying at the Faculty of Health Sciences of Bartın University. Students from each faculty to be included in the study were determined using a computer-assisted simple random sampling method. Students in the experimental and control groups were determined according to an algorithm created by a computer program called Research Randomizer. For the control group, 598 female students in İnönü University Nursing Department, numbers from 1 to 598 were randomly divided into a single set.For the experimental groups, 408 female students from the Faculty of Health Sciences of Bartın University were randomly divided into two sets (100 acupressure, 100 mindfulness), numbers numbered from 1 to 200. Which set will be acupressure and mindfulness group was determined by drawing lots. A research-independent academician made the selection blindly. As a result of the draw, it was determined that the first set was the acupressure group, and the second set was the mindfulness group. The assignment of the students to the experimental and control groups was made using the simple randomization method. Students were sorted by student number before randomization. Experimental and control groups were determined by the order given by the computer program Research Randomizer. The students who scored 110 and above were included in the study, after which the PMSS scale was applied to the determined students. In the study, it was accepted that 338 students who scored 110 and above from the scale experienced PMS. In the study, data were collected with the Participant Information Form, PMSS and WHOQOL-BREF. The acupressure group was asked to apply acupressure two days a week for 12 weeks, a total of 24 times. In the mindfulness group, 8 weeks of Conscious Awareness Stress Reduction Program was applied, after which the students were asked to practice mindfulness for 3 cycles. Students in both experimental groups were asked to stop the practices after acupressure and mindfulness practices. PMSS and WHOQOL-BREF were applied to both experimental and control groups as an intermediate test 12 weeks after the pre-test and a post-test 24 weeks later.

ELIGIBILITY:
Inclusion criteria

* Regular menstruation (between 21-35 days), being over 18 years old,
* Being single,
* Not using analgesics during menstruation,
* Not having any psychiatric diagnosis or gynecological disease (abnormal uterine bleeding, uterine fibroids, ovarian cysts, etc.),
* Not using contraceptives,
* Not having tissue deformities in the extremities and not having any health problems that can prevent physical exercise,
* A score of >110 on the PMSS scale.

Exclusion criteria

* Not participating in at least two mindfulness groups,
* Not having regular menstruation in the last 3 months,
* It is the use of analgesics during menstruation during the period of participating in the research.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 270 (Actual)
Dates: Start 2022-03-31 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
The Premenstrual Syndrome Scale (PMSS) | 6 month
  The scale consists of 44 questions. The lowest score that can be obtained from the scale is 44, and the highest score is 220. An increase in the score obtained from the scale indicates that the intensity of PMS symptoms increases. A total score above 110 in the premenstrual syndrome scale indicates the presence of PMS.

SECONDARY OUTCOMES:
The World Health Organization Quality of Life Assessment Questionnaire | 6 month
  On a five-point Likert-type scale, each
  A question is scored from 1 to 5, and a score can be obtained from 0-100 from the scale. An increase in the scores obtained from the scale indicates that the quality of life increases. While calculating the score of the scale, the 1st and 2nd questions are evaluated independently. In the calculation, the answers obtained from questions 3, 4, 26 and 27 are calculated by reversing. Since the scale does not have a total score, its sub-dimensions are used to evaluate the quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Simge ÖZTÜRK, PHD.Student, Study Chair — T.R. İNÖNÜ UNIVERSITY SCIENTIFIC RESEARCH AND PUBLICATION ETHICS COMMITTEE 2022/3172; Sermin TİMUR TAŞHAN, professor, Study Director — T.R. İNÖNÜ UNIVERSITY
Locations (1):
- Simge OZTURK, Malatya, Centre, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No